CLINICAL TRIAL: NCT03857724
Title: Clinical and Three-dimensional Ultrasound Assessment of Cases With Apical Prolapse Surgeries. A Prospective Cohort Study
Brief Title: Three-dimensional Ultrasound Assessment in Cases of Prolapse Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Yacoub Shafeek, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3D ULTRASOUND
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prolapse surgery (Experimental)
  Interventions: Procedure: prolapse surgery

INTERVENTIONS:
Procedure: prolapse surgery — prolapse surgery

SUMMARY:
The levator ani muscle seems to play a key role in pelvic floor dysfunction. This muscle has two major components, the pubovisceral (including the pubococcygeus and puborectalis muscles) and the iliococcygeal muscles.Major levator ani defects are associated with pelvic organ prolapse (POP) and POP recurrence

DETAILED DESCRIPTION:
The aetiology of female pelvic organ prolapse (FPOP) is complex and likely due to a combination of factors. Genetics, race, aging and menopause, obesity and conditions associated with a chronically increased intra-abdominal pressure such as chronic obstructive pulmonary disease as well as childbirth trauma have been implicated. Delivery-related trauma to the pubovisceral muscle is common and obviously associated with female pelvic organ prolapse.

It is a common problem with an incidence as high as 40%, and 10-20% of women will require surgery for prolapse at least once in their lifetime.

The levator hiatus defines the 'hernial portal' through which FPOP develops. Childbirth clearly leads to an enlargement of the levator hiatus, even in the absence of levator trauma.

And the levator hiatal dimensions are strongly associated with FPOP and with prolapse recurrence Enlargement of the levator hiatus is more likely to be the cause rather than the effect of FPOP. Alterations of the levator hiatus morphology following delivery have been demonstrated using magnetic resonance imaging (MRI) and more recently, three-dimensional (3D) ultrasound imaging Magnetic resonance imaging (MRI) has been shown to visualize levator ani defects effectively, but in recent years, translabial 3- and 4-dimensional (3D/4D) ultrasound has shown to provide valuable information on biometrical properties of the pelvic floor and morphology of the levator ani muscle.And recently three-dimensional ultrasonography is an alternative for MRI in detecting levator defects.

Currently, technologic advances in 3D ultrasonography allow access to the arbitrarily defined planes anywhere within ultrasound volume data and permit direct imaging of the entire levator hiatus.

Translabial three-dimensional ultrasonography has practical advantages because it is less expensive, easily accessible, and more readily available for gynecologists.

3D-Ultrasound in urogynecology could be helpful in diagnosing of urinary incontinence and urethral hypermobility, to document pelvic floor anatomy and to assess anatomic and functional changes before and after gynecologic surgery.

The objective of our research was to detect levator ani defects in women with POP before and after apical prolapse surgeries and if they will be corrected after the operation or not.

The secondary objective was to 1)detect the most appropriate surgical procedure in restoring the dimensions of the hiatal area.

2)Correlate between the levator ani defects and the complains, quality of life questionnaires, clinical examination of the patient before and after the surgery.

3)The role of 3D-Ultrasound in diagnosing the pelvic floor defects and targeting the Surgical procedure to restore the defects.

4)Introduce and stress on POP-Q system into Assuit general hospital and Abuteeg Hospital as it will be used to evaluate all cases both pre-operatively and during post-operative follow up being the standard method for evaluating cases of pelvic organ prolapse.

Objective cure was defined as the: absence of the prolapse as indicated by a POP-Q stage of 0-1.

ELIGIBILITY:
Inclusion Criteria:

I. Arabic female that is able to understand the instructions and the questionnaires that will be given II. Apical prolapse Stage 2-4 (according to POP-Q)(30,33) III. Sexually active (at least 3 times every month)

Exclusion Criteria:

1. Pregnancy
2. Postpartum women during the 1st 6 months postpartum
3. Human papillomavirus vulvar disease (condyloma acuminata)
4. Patient unfit for surgery
5. Previous pelvic reconstruction surgery.
6. Factors affecting healing process as uncontrolled diabetes, steroid therapy, on chemotherapy,….. etc

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
levator hiatus area in cm2 in women with POP before and after apical prolapse surgeries. | 2 years
  levator hiatus area in cm2 in women with POP before and after apical prolapse surgeries.

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital, Asyut, Egypt

REFERENCES:
- [Result] Rinne KM, Kirkinen PP. What predisposes young women to genital prolapse? Eur J Obstet Gynecol Reprod Biol. 1999 May;84(1):23-5. doi: 10.1016/s0301-2115(99)00002-0. PMID 10413222
- [Result] Lin KL, Juan YS, Chou SH, Long CY. Ultrasonographic Assessment with Three-Dimensional Mode of the Urethral Compression Effect following Sling Surgery with and without Mesh Surgery. Biomed Res Int. 2019 Jan 6;2019:8285351. doi: 10.1155/2019/8285351. eCollection 2019. PMID 30723744